CLINICAL TRIAL: NCT06449040
Title: Treatment of Cutaneous Leishmaniasis With Liposomal Amphotericin B in the Elderly: a Randomized Clinical Trial
Brief Title: Treatment of Cutaneous Leishmaniasis With Liposomal Amphotericin B in the Elderly
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Instituto Gonçalo Muniz FIOCRUZ BA (Unknown)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, Head of Immunology Service, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AmL Eld
Record Dates: First submitted 2024-05-28; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cutaneous Leishmaniasis, American
Keywords: Cutaneous Leishmaniasis; Liposomal Amphotericn B; L. braziliensis; Elderly
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis, Cutaneous | interventions — liposomal amphotericin B

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Anfo12mg/kg (Active Comparator): Liposomal amphotericin B (AmBisome®) - 3mg/kg twice a week; total dose of 12 mg/kg
  Interventions: Drug: Liposomal amphotericin B (AmBisome®)
- Group Anfo18mg/kg (Active Comparator): Liposomal amphotericin B (AmBisome®) - 3mg/kg twice a week; total dose of 18 mg/kg
  Interventions: Drug: Liposomal amphotericin B (AmBisome®)
- Group Anfo24mg/kg (Active Comparator): Liposomal amphotericin B (AmBisome®) - 3mg/kg twice a week; total dose of 24 mg/kg
  Interventions: Drug: Liposomal amphotericin B (AmBisome®)

INTERVENTIONS:
Drug: Liposomal amphotericin B (AmBisome®) — Liposomal amphotericin B (AmBisome®) - intravenous use, twice a week until total dose is achieved

SUMMARY:
A randomized controlled pilot trial with the aim of identifying the dose of liposomal amphotericin B associated with the highest cure rate in Cutaneous Leishmaniasis (CL). We selected 28 patients of both sexes, aged 60 years or older, diagnosed with CL and confirmed by detection of L. braziliensis DNA. The groups were treated with different total doses of medication: G1: 12 mg/kg; G2: 18mg/kg; G3: 24 mg/kg. Clinical and laboratory evaluations were carried out during the period of 180 days (D0, D15, D30, D60, D120, D150 and D180).

DETAILED DESCRIPTION:
The study was carried out through a randomized and double-blind pilot clinical trial, with the inclusion of patients treated at the Corte de Pedra Health Center, endemic region for Cutaneous Leishmaniasis. Twenty-eight patients participated in the study, after accepting and signing the Free and Informed Consent Form they were randomized through the list generated electronically by the website www.randomization.com and allocated into three groups.

The groups were treated with liposomal amphotericin B (AmBisome®) with three different total doses: Group 1 (G1) total dose of 12 mg/kg (10 patients). Group 2 (G2): 18 mg/kg (9 patients). Group 3 (G3): 24 mg/kg (9 patients). The drug was used twice a week in a hospital outpatient setting. Clinical evaluations were performed before starting therapy (D0), and at D15, D30, D60, D120 and D180. Laboratory evaluations (hemogram, BUN, Creatinine, K, ALT, AST) were determined on D0, D15 and D30 or D60.

ELIGIBILITY:
Inclusion Criteria:

* CL clinical diagnosis (presence of an ulcer)
* CL confirmed by detection of amastigotes in pathology and/or positive PCR for L. braziliensis in tissue obtained from the ulcer border
* Presence of one to a maximum of three ulcers
* Ulcer size between 1 and 5 mm
* Ulcer evolution of 1 to 6 months

Exclusion Criteria:

* Previous CL treatment
* Renal or hepatic disease
* HIV co-infection.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Total initial cicatrization | 30 to 90 days after the first day of treatment
  Healing of the total ulcer area, without elevation of the ulcer edges upon clinical evaluation

SECONDARY OUTCOMES:
Total final cicatrization | 30 to 180 days after the first day of treatment
  Healing of the total ulcer area, without elevation of the ulcer edges upon clinical evaluation
Time to cure | 30 to 180 days after the first day of treatment
  Number of days from the first day of treatment until total ulcer cicatrization

CONTACTS AND LOCATIONS:
Overall Officials: PAULO MACHADO, MD, PhD, Principal Investigator — Federal University of Bahia
Locations (1):
- Corte de Pedra Health Post, Presidente Tancredo Neves, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No